CLINICAL TRIAL: NCT01934244
Title: Evaluation of the Safety of NovaSure in the Presence of Essure Following the Essure Confirmation Test (ECT) Post-Approval Study
Brief Title: Post Approval NovaSure Essure Labeling Study
Acronym: PANEL
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: S0112003
Record Dates: First submitted 2013-08-26; First posted 2013-09-04 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Menorrhagia
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Per Protocol: All enrolled patients in which all inclusion/exclusion criteria were met and the NovaSure endometrial ablation was completed.
  Interventions: Device: NovaSure Endometrial Ablation
- Primary: All enrolled patients in whom the Novasure device was inserted.
- Intent to treat: All enrolled patients in which NovaSure device was attempted.

INTERVENTIONS:
Device: NovaSure Endometrial Ablation — The NovaSure Endometrial Ablation device consists of a disposable single-use, conformable bipolar electrode array mounted on an expandable frame that can create a confluent lesion on the entire interior surface area of the uterine cavity. The device is inserted transcervically into the uterine cavity, and the sheath is retracted to allow the bipolar electrode array to be deployed and conform to the uterine cavity. The disposable device works in conjunction with a dedicated NovaSure RF (radio frequency) controller to perform customized, global endometrial ablation.
  Groups: Per Protocol

SUMMARY:
This post approval, observational study is being conducted to further evaluate the safety of the NovaSure Endometrial Ablation System when it is performed in the presence of Essure micro-inserts.

DETAILED DESCRIPTION:
A prospective, single arm, multi-center, post approval study that is designed to provide additional information on the safety of performing a NovaSure Impedence Controlled Endometrial Ablation System in the presence of Essure Permanent Birth Control System, following the Essure Confirmation Test has confirmed both bilateral tubal occlusion and the satisfactory location of the Essure micro-inserts. The study will be conducted at up to 15 clinical sites and enroll 318 patients. Patients who meet the inclusion and none of the exclusion criteria will have the study explained to them and be invited to participate. Enrolled subjects will have baseline data collected at the time of their NovaSure procedure and will be followed for 1 month after the NovaSure procedure to be assessed for adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older and premenopausal.
* Subject's gynecological history supports the use of NovaSure endometrial ablation for the treatment of menorrhagia.
* Subject has had an Essure Permanent Birth Control System procedure.
* The Essure Confirmation Test has confirmed both bilateral tubal occlusion and satisfactory placement of the Essure micro-inserts. A written report or ECT radiologic films need to be provided by the physician who performed the ECT. If neither is available, the ECT must be repeated prior to enrollment.
* Subject is able to provide informed consent

Exclusion Criteria:

* Subject has known or suspected endometrial carcinoma (uterine cancer) or pre-malignant conditions of the endometrium, such as unresolved (atypical) adenomatous hyperplasia.
* Subject has abnormal/obstructive uterine cavity as confirmed by hysteroscopy or other imaging study (e.g. congenital malformation, large fibroid or large polyp)
* Subject with any anatomic condition (e.g. history of previous classical cesarean section or transmural myomectomy) or pathologic condition (e.g. long term medical therapy) that could lead to weakening of the myometrium.
* Subject has an active genital or urinary tract infection at the time of the procedure (e.g., cervicitis, vaginitis, endometritis, salpingitis, or cystitis).
* Subject has an intrauterine device (IUD) currently in place.
* Subject has active pelvic inflammatory disease or history of recent pelvic infection.
* Subject has undiagnosed vaginal bleeding.
* ECT unable to adequately assess bilateral tubal occlusion and proper micro-insert placement.
* Subject has uterine sound measurement greater than 10 cm.
* Subject with a uterine cavity length less than 4 cm.
* Subject with a uterine cavity width less than 2.5 cm, as determined by the width dial of the disposable NovaSure device following device deployment.
* Subject is unable to comply with the protocol and be available for follow up
* In the opinion of the investigator, the subject has a medical condition that precludes safe participation in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Premenopausal women 18 years of age or older who have abnormal uterine bleeding and are candidates for a NovaSure Endometrial Ablation that have already had an Essure Permanent Birth Control system procedure and an Essure Confirmation Test that has confirmed both bilateral tubal occlusion and the satisfactory location of the Essure micro-inserts.
Sampling Method: Non-Probability Sample
Enrollment: 318 (Estimated)
Dates: Start 2013-12 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Essure micro-insert removal with NovaSure device | NovaSure procedure visit (Day 1)
  At the end of the NovaSure treatment and upon removal of the NovaSure device, the device will be directly observed to see if any Essure micro-insert(s) is(are) attached.

SECONDARY OUTCOMES:
Number and percentage of subjects with adverse events | NovaSure Procedure visit (Day 1) and 1 month post NovaSure procedure
  Adverse events reported during and/or immediately post operative the NovaSure procedure.
  Adverse events reported up to 1 month after the NovaSure procedure

CONTACTS AND LOCATIONS:
Overall Officials: Edward Evantash, MD, Study Director — Hologic, Inc.
Locations (14):
- United States (14):
  - New Horizon Women's Care, Chandler, Arizona
  - Westside Women's Care, Arvada, Colorado
  - Physicians Care Clinical Research, LLC, Sarasota, Florida
  - Western DuPage Obstetrics and Gynecology, Downers Grove, Illinois
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Saginaw Valley Medical Research Group, LLC, Saginaw, Michigan
  - Minnesota Gynecology and Surgery, Edina, Minnesota
  - Bosque Women's Care, Albuquerque, New Mexico
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Seven Hills Women's Center, Cincinnati, Ohio
  - Amy Brenner MD & Associates, LLC, West Chester, Ohio
  - Chattanooga Medical Research, LLC, Chattanooga, Tennessee
  - Tennessee Women's Care, Nashville, Tennessee
  - Rockwood Clinic, P.S., Spokane, Washington

REFERENCES:
- [Background] Basinski CM, Price P, Burkhart J, Johnson J. Safety and Effectiveness of NovaSure(R) Endometrial Ablation After Placement of Essure(R) Micro-Inserts. J Gynecol Surg. 2012 Apr;28(2):83-88. doi: 10.1089/gyn.2011.0061. PMID 24761128
- [Background] Saunders, D: Essure and Endometrial Ablation: Clinical studies and case reviews of Essure with 118 NovaSure procedures, Supplement to OBG Management, April, 2010.
- See also: Hologic, Inc. website — http://www.hologic.com